CLINICAL TRIAL: NCT05433662
Title: Pandemic Acceptance and Commitment Therapy (Pan-ACT): Feasibility and Acceptability of Telehealth Delivery With Older Veterans
Brief Title: Telehealth Acceptance and Commitment Therapy for Older Veterans Experiencing Pandemic-Related Stress
Acronym: Pan-ACT
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Other Study IDs: D3898-P; 1I21RX003898-01A1 (NIH)
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Psychological Stress
Keywords: Older adult; acceptance and commitment therapy; telehealth; pandemic
MeSH Terms: conditions — Stress, Psychological | interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Veterans: Veterans will be ages 65 and older, cognitively intact, and experiencing pandemic-related stress.
  Interventions: Behavioral: Pandemic Acceptance and Commitment Therapy (Pan-ACT)

INTERVENTIONS:
Behavioral: Pandemic Acceptance and Commitment Therapy (Pan-ACT) — Pan-ACT is a 10-session, closed group, transdiagnostic intervention for older adults.
  Other Names: Acceptance and Commitment Therapy (ACT); ACT for Older Adults; The Third ACT

SUMMARY:
Older adults have been disproportionately impacted and distressed by the COVID-19 pandemic. Social distancing and stay-at-home orders have increased older adults' risk of social isolation and loneliness that will has led to a pandemic-induced fear of being in close proximity to other people. These fears and avoidant behaviors will have lasting effects if not treated with effective, safe, and convenient psychological interventions. This study will evaluate the acceptability and feasibility of delivering a small group intervention, called Acceptance and Commitment Therapy (ACT), through a telehealth modality to Veterans ages 65 and older who are experiencing pandemic-related emotional and physical distress. ACT helps decrease emotional suffering, improve well-being and promote positive behavior change by increasing one's psychological flexibility through the practice of mindfulness, acceptance, and values-based behaviors. The knowledge gained from this study will be used to better tailor the invention to meet the needs of older Veterans in an era of post-pandemic recovery.

DETAILED DESCRIPTION:
Significance: Accounting for over 80% of COVID-19 related deaths in the United States, adults ages 65 and older have been disproportionately impacted by this pandemic more than any other age group. As a result, they may bear a heavy psychological burden in the months and years to come. Older adults have been labeled "vulnerable" to COVID-19 and strongly encouraged to adhere to "social distancing." This prevention measure is meant to mitigate the spread of the virus but has increased older adults' risk of social isolation and loneliness, which are two known correlates of increased morbidity and mortality in late life. Pandemic-related restrictions have decreased older adults' life-space mobility and negatively affected their physical and nutritional well-being, impairing their quality of life and potentially increasing their vulnerability to poorer outcomes if exposed to COVID-19. Research has documented a plethora of pandemic-related stressors that are common among older adults (e.g., fear of infection, loss of loved ones, financial repercussions) and the culminating psychological impact. Telehealth-adapted evidence-based psychological interventions are needed to address the psychosocial and physical toll of the pandemic among older Veterans. Acceptance and Commitment Therapy (ACT) decreases emotional suffering, improves well-being, promotes and supports healthy behavior changes, and treats a wide range of diagnoses by increasing psychological flexibility through mindfulness, acceptance, and values-based behaviors. Higher psychological flexibility has been associated with pandemic-related coping and well-being. Randomized studies of ACT with older adults are few but promising, and most research studies with this population have used a group format. While research on telehealth delivery of ACT for older adults is limited, preliminary results indicate it is feasible and as effective as ACT delivered in person.

Specific Aim: The proposed study will pilot a 10-session telehealth Pandemic ACT group intervention (i.e., Pan-ACT group) with Veterans ages 65 and older who are experiencing pandemic-related emotional and physical distress.

Methods and Procedures: Twenty-five older Veterans will be enrolled in this single-arm feasibility pilot trial. The intervention will be delivered weekly in 90-minute sessions of groups of four to five Veterans. Feasibility and acceptability of study procedures will be measured by referred-to-enrolled rate, telehealth access and capability, electronic data collection of outcome measures, and qualitative feedback on data collection procedures and measures. Feasibility and acceptability of the intervention will be measured by attendance; attrition; homework completion; participant ratings of the intervention's feasibility, acceptability, and fit; qualitative feedback; and treatment fidelity. Preliminary responsiveness of outcomes measures will be explored. Participants will complete measures of pandemic-related emotional and physical distress, psychological flexibility, depression, anxiety, social connectedness, perceived health, functional impairment, and meaningful engagement at baseline, posttreatment, and one-month follow-up. A brief midpoint assessment at week 5 of the group will consist of measures of social connectedness and functional impairment. Qualitative data will be gathered on perceived efficacy to implement intervention skills and specific emotional or behavioral changes participants have noticed in themselves as a result of the intervention.

Conclusion: The telehealth Pan-ACT Group is a mental and behavioral health rehabilitation intervention that focuses on helping older Veterans develop or recover coping skills that were lost or are no longer effective during the ongoing COVID-19 pandemic. The proposed study address a major research and clinical gap by gathering new knowledge for an urgent need, which will inform the development of a full-scale randomized controlled trial to evaluate the intervention's effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* receives care at Tuscaloosa VA Medical Center
* score of 9 or greater on the COVID-19 Mental Health Impacts Scale
* English speaking
* provides written informed consent

Exclusion Criteria:

* diagnosis of dementia
* score of 31 or less on the Modified Telephone Interview for Cognitive Status
* actively suicidal or homicidal
* actively psychotic
* unstable medical condition
* active substance use disorder
* currently participating in another CBT-based intervention

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans ages 50 and older receiving services at the Tuscaloosa VA Medical Center (TVAMC) will be recruited from primary care, home-based primary care, and mental health clinics.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Acceptability of study protocol - retention | Through study completion, approximately 2 years
  Rate of study completion
Feasibility of study protocol - telehealth | Through study completion, approximately 2 years
  Percent of participants who have telehealth capability for duration of intervention
Acceptability of intervention - group attendance | Through study completion, approximately 2 years
  Percent of participants who attend 70% or more of intervention sessions

OTHER OUTCOMES:
Acceptability of study protocol - enrollment | Throughout active enrollment period, approximately 1.5 years
  Referred to enrolled rate
Acceptability of study protocol - assessment completion | Through study completion, approximately 2 years
  Rate of completed study assessments
Feasibility of study protocol - timeline | Through study completion, approximately 2 years
  Percent of group cohorts that start as scheduled on timeline
Acceptability of intervention - homework completion | Through study completion, approximately 2 years
  Percent of completed home practice exercises
Feasibility of intervention - treatment fidelity | Through study completion, approximately 2 years
  Ratings on ACT Fidelity Measures

CONTACTS AND LOCATIONS:
Overall Officials: Lori Lynne Davis, MD AB, Principal Investigator — Tuscaloosa VA Medical Center, Tuscaloosa, AL
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Data sets will have no identifying information of participants (participants ages above 89 will be coded as "90 or above" in accordance with HIPAA regulations). In addition, no Clinical Site identifiers beyond the code numbers will be included in the data set. A "dictionary" dataset will also be included which will include description labels for all the variables. The archives will also include the data collection forms and data collection instructions, including coding schemes and scoring algorithms, and study manuals. These documents will be archived as Adobe Acrobat (.pdf) files. No audio files, video files, or qualitative transcripts will be shared.

DOCUMENTS (1):
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT05433662/ICF_000.pdf